CLINICAL TRIAL: NCT01421134
Title: A Randomized, 6-Week, Double-Blind, Placebo-Controlled, Flexible-Dose, Parallel-Group Study of Lurasidone for the Treatment of Major Depressive Disorder With Mixed Features
Brief Title: Major Depressive Disorder (MDD) With Mixed Features - Flexible Dose
Acronym: RESOLVE 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1050304
Record Dates: First submitted 2011-08-17; First posted 2011-08-22 (Estimated); Results first posted 2015-10-09 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Major Depressive Disorder With Mixed Features
Keywords: depression; Lurasidone; Latuda
MeSH Terms: conditions — Depression | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lurasidone (Experimental): Lurasidone 20, 40 or 60 mg
  Interventions: Drug: Lurasidone
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lurasidone — 20, 40, 60 mg, flexible dose, once daily PM 6 weeks
  Other Names: Latuda
  Arms: Lurasidone
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Lurasidone HCl is a compound that is a candidate for the treatment of major depressive with mixed features.This clinical study is designed to test how well Lurasidone works to treat major depressive disorder with mixed features.

ELIGIBILITY:
Inclusion Criteria:

* Subject provides written informed consent and is willing and able to comply with the protocol in the opinion of the Investigator.
* Subject is 18 to 75 years of age, inclusive.
* Subject has MDD (diagnosed by DSM-IV-TR, and confirmed by the Structured - Clinical Interview for DSM-IV Disorders - Clinical Trial version [SCID-CT]).
* Subject is currently experiencing a major depressive episode (diagnosed by DSM IV TR; at least 2 weeks in duration) AND two or three of the following manic symptoms occurring on most days over at least the last 2 weeks (confirmed by the SCID-CT modified for Study D1050304):

  * Elevated, expansive mood
  * Inflated self-esteem or grandiosity
  * More talkative than usual or pressure to keep talking
  * Flight of ideas or subjective experience that thoughts are racing
  * Increase in energy or goal-directed activity (either socially, at work or school, or sexually)
  * Increased or excessive involvement in activities that have a high potential for painful consequences (e.g., engaging in unrestrained buying sprees, sexual indiscretions, or foolish business investments)
  * Decreased need for sleep (feeling rested despite sleeping less than usual; to be contrasted from insomnia)

Exclusion Criteria:

* Subject has Axis I or Axis II diagnosis other than MDD that has been the primary focus of treatment within the 3 months prior to screening.
* Subject answers "yes" to "Suicidal Ideation" Item 4 or 5 on the C-SSRS (at time of evaluation) at screening or baseline visit.
* Subject has attempted suicide within the past 3 months.
* Subject has a lifetime history of any bipolar I manic or mixed manic episode.
* Subject has any abnormal laboratory parameter at screening that indicates a clinically significant medical condition as determined by the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2011-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (43):
- United States (19):
  - Birmingham Psychiatry Pharmaceutical Studies, Inc., Birmingham, Alabama
  - Synergy Clinical Research Center, Escondido, California
  - Collaborative Neuroscience Network Inc., Garden Grove, California
  - Stanford -VA Palo Alto Health Care System, Palo Alto, California
  - Clinical Innovations Inc., Riverside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Florida Clinical Research Center, LLC, Sarasota, Florida
  - Massachusetts General Hospital - Center for Anxiety and Traumatic Stress Disorders, Boston, Massachusetts
  - St. Charles Psychiatric Associates/Midwest Research Group, Saint Charles, Missouri
  - Social Psychiatric Research Inst. (SPRI) Clinical Trials, Brooklyn, New York
  - Village Clinical Research Inc., New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Behavioral Medical Research of Staten Island, Staten Island, New York
  - Psychiatry and Behavioral Sciences, Duke, Durham, North Carolina
  - Midwest Clinical Research Center, Dayton, Ohio
  - CRI Worldwide - Kirkbride, Philadelphia, Pennsylvania
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Dept. of Psychiatry, UT Southwestern Medical Center, Dallas, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
- Russia (6):
  - Saint Nicholas Psychiatric Hospital., Saint Petersburg
  - City Psychiatry Hospital 4 (Saint Petersburg Psychiatric Admitting Unit), Saint Petersburg
  - Federal State Institution "Saint-Petersburg Research psychoneurogical Institute named after V.M. Bekhtereva", Saint Petersburg
  - Municipal Healthcare Institution"City Clinical Hospital #2, n.a. V.I. Razumovsky" of Healthcare Committee of Administration of Municipal Entity "City of Saratov", Saratov
  - State Healthcare Institution, Saratov Regional Psychiatric Hospital of St.Sophia,, Saratov
  - Limited Liability Company "Research-And-Educational Centre of Psychotherapy "Podderzhka", Stavropol
- Serbia (9):
  - Institute of Mental Health, Belgrade
  - Psychiatric Clinic, Clinical Hospital Center"Dr. Dragisa Misovic-Dedinje", Belgrade
  - Health Centre Cacak Department of Psychiatry, Čačak
  - Clinical Center Nis, Psychiatric Clinic, Gornja Toponica
  - Clinical Center Kragujevac, Psychiatric Clinic, Kragujevac
  - Clinic for Mental Health, Clinical Center Nis, Niš
  - Special Hospital for Psychiatric Diseases "Sveti Vracevi", Vojvodina
  - Special Hospital for Psychiatric Diseases "Dr Slavoljub Bakalovic", Vršac
  - General Hospital "Djordje Joanovic" Psychiatric Dept., Zrenjanin
- Ukraine (7):
  - Dnipropetrovsk Regional Clinical Hospital named Mechnikov, Dnipropetrovsk
  - State Institution "Institute of Neurology, Psychiatry and Narcology NAMS of Ukraine", Dep. of Clinical, Social and Child Psychiatry, Kharkiv
  - Communal Institution of Kyiv Regional Council "Regional Psychiatric and Narcological Medical Association "Psychiatric Dept. #10 and Psychiatric Dept. #2, Kyiv
  - "Lugansk State Medical University"Chair of Psychiatry, Narcology and Medical Psychology; Lugansk Regional Clinical Psychoneurological Hospital, Dispensary Dept. for adults, Luhansk
  - Municipal Institution "Lviv Regional State Clinical Psychiatric Hospital, Department #20, Lviv
  - Odesa Regional Psychoneurological Dispensary, Outpatient Dept., Odesa
  - Vinnytsya National Medical University n.a. M.I. Pyrogov, Dept. of Psychiatry and Narcology, Vinnytsya Regional Psychoneurological Hospital n.a. O.I. Yushchenko, Dept. no. 14, Dept. no 15, Vinnytsia
- United Kingdom (2):
  - MAC Clinical Research Limited, Cannock
  - MAC Clinical Research Limited, Manchester

REFERENCES:
- [Derived] Clayton AH, Tsai J, Mao Y, Pikalov A, Loebel A. Effect of Lurasidone on Sexual Function in Major Depressive Disorder Patients With Subthreshold Hypomanic Symptoms (Mixed Features): Results From a Placebo-Controlled Trial. J Clin Psychiatry. 2018 Aug 7;79(5):18m12132. doi: 10.4088/JCP.18m12132. PMID 30086213
- [Derived] Targum SD, Pendergrass JC, Lee S, Loebel A. Ratings surveillance and reliability in a study of major depressive disorder with subthreshold hypomania (mixed features). Int J Methods Psychiatr Res. 2018 Dec;27(4):e1729. doi: 10.1002/mpr.1729. Epub 2018 Jun 26. PMID 29943445
- [Derived] Targum SD, Suppes T, Pendergrass JC, Lee S, Silva R, Cucchiaro J, Loebel A. Major depressive disorder with subthreshold hypomania (mixed features): Clinical characteristics of patients entered in a multiregional, placebo-controlled study. Prog Neuropsychopharmacol Biol Psychiatry. 2016 Jul 4;68:9-14. doi: 10.1016/j.pnpbp.2016.02.007. Epub 2016 Feb 22. PMID 26908089

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lurasidone | Placebo
Started | 109 | 102
Completed | 102 | 87
Not Completed | 7 | 15
Not completed — Adverse Event | 3 | 5
Not completed — Lack of Efficacy | 2 | 4
Not completed — Protocol Violation | 0 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Administrative | 0 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Two subjects were randomized in error and were not treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lurasidone | Placebo | Total
Number analyzed (Participants) | 109 | 100 | 209
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 106 | 96 | 202
  >=65 years | 2 | 4 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (12.08) | 46.4 (12.01) | 44.9 (12.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 72 | 145
  Male | 36 | 28 | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 12 | 26
  White | 94 | 86 | 180
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Russian Federation | 18 | 13 | 31
  United States | 34 | 26 | 60
  Ukraine | 30 | 32 | 62
  United Kingdom | 1 | 3 | 4
  Serbia | 26 | 26 | 52

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to the 6-week Study Endpoint in Montgomery-Asberg Depression Rating Scale (MADRS) Total Scores
Description: The MADRS consists of 10 items, each rated on a Likert scale, from 0="Normal" to 6="Most Severe". The MADRS total score is calculated as the sum of the 10 items. The MADRS total score ranges from 0 to 60. Higher scores are associated with greater severity.
Time Frame: Baseline to Week 6
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone | Placebo
Number analyzed (Participants) | 108 | 100
units on a scale | -20.5 (0.95) | -13.0 (1.00)
Statistical Analysis 1: Comparison: Lurasidone vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Least Square Mean Difference = -7.5, 95% CI 2-sided [-10.2 to -4.8], Standard Error of Mean 1.37

2. Secondary Outcome: Mean Change From Baseline to the 6-week Study Endpoint in the Clinical Global Impression-Severity of Illness (CGI-S) Score
Description: The CGI-S score is a single value, clinician-rated assessment of illness severity and ranges from 1= 'Normal, not at all ill' to 7= 'Among the most extremely ill patients'. A higher score is associated with greater illness severity.
Time Frame: Baseline to Week 6
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone | Placebo
Number analyzed (Participants) | 108 | 100
units on a scale | -1.83 (0.109) | -1.18 (0.115)
Statistical Analysis 1: Comparison: Lurasidone vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Least Square Mean Difference = -0.65, 95% CI 2-sided [-0.96 to -0.34], Standard Error of Mean 0.157

3. Secondary Outcome: Mean Change From Baseline to Week 6 in the Young Mania Rating Scale (YMRS) Total Score
Description: The YMRS is an 11-item clinician-rated instrument used to assess the severity of mania. Seven items are rated on a 5-point scale, ranging from 0 to 4, and four items are rated on a 9-point scale, ranging from 0 to 8. The YMRS total score is calculated as the sum of the 11 individual items and ranges from 0 to 60. Higher scores are associated with greater severity of mania.
Time Frame: Baseline to Week 6
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone | Placebo
Number analyzed (Participants) | 108 | 100
units on a scale | -7.0 (0.35) | -4.9 (0.37)
Statistical Analysis 1: Comparison: Lurasidone vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Least Square Mean Difference = -2.1, 95% CI 2-sided [-3.1 to -1.1], Standard Error of Mean 0.50

4. Secondary Outcome: Mean Change From Baseline to Week 6 in the Sheehan Disability Scale (SDS) Total Score
Description: The SDS is a composite of three self-rated items designed to measure the extent to which three major sectors (work/school, social life/leisure, and family life/home responsibility) in the patient's life are impaired by depressive symptoms. These three items are responded to on a visual analogue scale (VAS) ranging through 0 (no impairment), 1-3 (mild), 4-6 (moderate), 7-9 (marked) and 10 (extreme) disability. The SDS total score is calculated as the sum of the three items and ranges from 0 (unimpaired) to 30 (highly impaired).
Time Frame: Baseline to Week 6
Population: Intent to treat population: If a subject has not worked/studied at all during the past week for reasons unrelated to the disorder, the SDS total score will be set to missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone | Placebo
Number analyzed (Participants) | 70 | 69
units on a scale | -11.2 (0.88) | -6.4 (0.88)
Statistical Analysis 1: Comparison: Lurasidone vs Placebo; Test type: Superiority or Other; p = 0.0001, ANCOVA; Least Square Mean Difference = -4.8, 95% CI 2-sided [-7.2 to -2.4], Standard Error of Mean 1.21

5. Secondary Outcome: Mean Change From Baseline to Week 6 in the Hamilton Rating Scale for Anxiety(HAM-A) Total Score
Description: The HAM-A is used to quantify the severity of anxiety symptomatology and consists of 14 items. Each item is rated on a 5-point scale, ranging from 0 (not present) to 4 (severe/disabling). The HAM-A total score is calculated as the sum of the 14 individual items and ranges from 0 to 56. Higher scores are associated with greater degree of anxiety.
Time Frame: Baseline to Week 6
Population: Intent to treat population. 3 Lurasidone subjects and 2 placebo subjects did not have post-baseline HAM-A assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone | Placebo
Number analyzed (Participants) | 105 | 98
units on a scale | -9.9 (0.58) | -5.4 (0.59)
Statistical Analysis 1: Comparison: Lurasidone vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Square Mean Difference = -4.5, 95% CI 2-sided [-6.1 to -2.9], Standard Error of Mean 0.81

6. Secondary Outcome: Percentage of Subjects Who Achieve a Response, Defined as ≥ 50% Reduction From Baseline on the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at Week 6 (LOCF).
Time Frame: Baseline to Week 6
Population: Intent to treat population
Measure: Number; unit: percentage of subjects
Arm/Group | Lurasidone | Placebo
Number analyzed (Participants) | 108 | 100
percentage of subjects | 64.8 | 30.0
Statistical Analysis 1: Comparison: Lurasidone vs Placebo; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 6.615, 95% CI 2-sided [3.251 to 13.459] — Odds Ratio was based on a logistic regression of response, with treatment group, baseline MADRS total score, and pooled center as fixed effects

7. Secondary Outcome: Percentage of Subjects Who Achieve a Remission, Defined as a Montgomery-Asberg Depression Rating Scale (MADRS) Total Score of ≤ 12 at Week 6 (LOCF)
Time Frame: Baseline to Week 6
Population: Intent to treat population
Measure: Number; unit: percentage of subjects
Arm/Group | Lurasidone | Placebo
Number analyzed (Participants) | 108 | 100
percentage of subjects | 49.1 | 23.0
Statistical Analysis 1: Comparison: Lurasidone vs Placebo; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 4.270, 95% CI 2-sided [2.105 to 8.663]

ADVERSE EVENTS:
Time Frame: 6 Weeks
Arm/Group | Lurasidone | Placebo
Serious Adverse Events (participants affected / at risk) | 1/109 | 0/100
Other Adverse Events (participants affected / at risk) | 31/109 | 29/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone (N=109) | Placebo (N=100)
Depression Suicidal (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone (N=109) | Placebo (N=100)
Nausea (Gastrointestinal disorders) | 7 (7) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 4 (5) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 2 (3)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 6 (6) | 6 (7)
Somnoelence (Nervous system disorders) | 5 (6) | 1 (1)
Akathisia (Nervous system disorders) | 4 (4) | 2 (2)
Dizziness (Nervous system disorders) | 4 (5) | 3 (3)
Insomnia (Psychiatric disorders) | 6 (7) | 11 (11)
Anxiety (Psychiatric disorders) | 4 (4) | 9 (12)
Haemarturia (Renal and urinary disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS agreement between Principal Investigator and Sponsor that restricts PI's rights to discuss or publish trial results after trial is completed.

In addition to the <60-180 day restriction above, since this is a multicenter study, 1st publication of study results shall be made with other participating study sites as a multicenter publication provided, if a multicenter publication is not forthcoming within 24 months post completion of study at all sites, PI shall be free to publish.